CLINICAL TRIAL: NCT02392533
Title: Ultrasound Confirmation of Neuraxial Anesthetic Vertebral Level in Post-partum Patients
Brief Title: Ultrasound and Neuraxial Anesthesia in Pregnancy
Acronym: USPREG
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB14-1556
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Infusion Site Anaesthesia
Keywords: ultrasound
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre cohort group: Following 3 months of data collection (pre-cohort group), education regarding the documented intervertebral space versus the actual intervertebral space that the neuraxial anesthetic was administered will be provided to each anesthesiologist and resident. Following delivery of this information, an additional 3 months of data collection will be performed (post-cohort group) (the same as the first 3 months) to evaluate whether a practice change took place.
  Interventions: Other: Education
- Post cohort group.: Following 3 months of data collection (pre-cohort group), education regarding the documented intervertebral space versus the actual intervertebral space that the neuraxial anesthetic was administered will be provided to each anesthesiologist and resident. Following delivery of this information, an additional 3 months of data collection will be performed (post-cohort group) (the same as the first 3 months) to evaluate whether a practice change took place.

INTERVENTIONS:
Other: Education — Education
  Groups: Pre cohort group

SUMMARY:
Ultrasonography is routinely performed during pregnancy by obstetricians to visualize the fetus, making patients familiar and comfortable with its usage. Ultrasonography does not result in adverse effects to the mother or fetus and is readily available at most facilities, yet is not routinely used to identify lumbar interspaces prior to providing neuraxial anesthesia. Ultrasonography is a valuable tool for accurately identifying lumbar intervertebral spaces and is more accurate than simple palpation of obscure anatomic landmarks. The investigators are interested to know the accuracy of anatomic landmark palpation in predicting the lumbar interspace of neuraxial anesthesia administration compared to identification of the interspace by ultrasound. The investigators are also interested in presenting anesthesia providers with feedback regarding their accuracy and then investigating whether this feedback causes a change in provider practice (i.e. use of ultrasound) or improved identification of the interspace prior to providing neuraxial anesthesia.

DETAILED DESCRIPTION:
Informed consent will be obtained and documented. All post-partum patients who received neuraxial anesthesia will be asked to provide consent for ultrasound to be used at their bedside to identify the interspace where the neuraxial anesthetic was administered. A low frequency ultrasound probe and sterile gel will be used to perform the less than five-minute study. The site of the neuraxial anesthetic placement will be identified by the puncture mark on the skin. The investigators will note the patient's medical record number and BMI, the names of the resident and attending anesthesiologist who placed the neuraxial anesthetic, the documented intervertebral space at the time of neuraxial anesthetic placement, anesthetic type, whether ultrasound was used for the initial neuraxial placement, and the documented intervertebral space identified post-partum by ultrasound.

Following 3 months of data collection, information regarding the documented intervertebral space versus the actual intervertebral space that the neuraxial anesthetic was administered will be provided to each anesthesiologist and resident. Following delivery of this information, an additional 3 months of data collection will be performed (the same as the first 3 months) to evaluate whether a practice change took place.

ELIGIBILITY:
Inclusion Criteria: All post-partum patients > 18 years old who had neuraxial anesthesia for delivery and are English Speaking.

-

Exclusion Criteria: Age < 18 years and non-English speaking, and did not have neuraxial anesthesia for delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-partum patients who had neuraxial anesthesia for their delivery.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Ultrasound identification of lumbar interspace | 3 months
  Number of vertebral levels different between lumbar interspace on palpation versus on ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Scavone, MD, Principal Investigator — The University of Chicago MEDICINE
Locations (1):
- The University of Chicago MEDICINE, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wallace DH, Currie JM, Gilstrap LC, Santos R. Indirect sonographic guidance for epidural anesthesia in obese pregnant patients. Reg Anesth. 1992 Jul-Aug;17(4):233-6. PMID 1515392
- [Result] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Result] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Efficacy of ultrasound imaging in obstetric epidural anesthesia. J Clin Anesth. 2002 May;14(3):169-75. doi: 10.1016/s0952-8180(01)00378-6. PMID 12031746
- [Result] Broadbent CR, Maxwell WB, Ferrie R, Wilson DJ, Gawne-Cain M, Russell R. Ability of anaesthetists to identify a marked lumbar interspace. Anaesthesia. 2000 Nov;55(11):1122-6. doi: 10.1046/j.1365-2044.2000.01547-4.x. PMID 11069342